CLINICAL TRIAL: NCT01027533
Title: Visual Performance of New Apodized Diffractive Multifocal IOL With Addition of Plus Three
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Marcony R Santhiago, University of São Paulo
Other Study IDs: MRS.1703
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2009-03

CONDITIONS: To Study the Influence of an Multifocal Intraocular Lens With Different Addition on Intermediate Visual Acuity
Keywords: multifocal intraocular lens; visual acuity; presbiopia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Restor +3: patients will be implanted bilaterally with Restor + 3
  Interventions: Other: Implantation of a multifocal Intraocular lens
- restor +4: Patients will be implanted bilaterally with Restor +4
  Interventions: Other: Implantation of a multifocal Intraocular lens

INTERVENTIONS:
Other: Implantation of a multifocal Intraocular lens — Bilateral implantation of a multifocal IOl
  Other Names: Restor + 3 SN6AD1; Restor + 4 SN6AD3

SUMMARY:
The purpose of the study is to determine whether implantation of a multifocal IOL with a modified addition at lens plane(Restor +3) results in better intermediate visual acuity with similar performance at distance and near compared to other multifocal IOL with similar design but with higher addition at lens plane. Patient's contrast sensitivity of vision and best reading distance following Restor +3 implantation were also assessed.

Study hypothesis: the implantation of an intraocular lens (IOL) with a modified addition at lens plane (restor +3, Alcon Laboratories,Inc) results in better intermediate visual acuity with similar distance and near visual acuity after cataract surgery.

DETAILED DESCRIPTION:
Patients with bilateral visually significant cataract with corneal astigmatism lower than 1.0D (diopters) will be eligible for inclusion in the study. Exclusion criteria will be any ocular diseases, such as corneal opacities or irregularity, dry eye, amblyopia, anisometropia, glaucoma, retinal abnormalities, surgical complications, IOL tilt, IOL decentration greater than 0.4 mm (estimated by retroillumination), or incomplete follow-up.

Patients will be examined before surgery and at 1, 7, 30, 90 days and 3and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* •Patients with bilateral visually significant cataract with corneal astigmatism lower than 1.0D (diopters)

Exclusion Criteria:

* Ocular diseases, such as corneal opacities or irregularity, dry eye amblyopia, anisometropia, glaucoma, retinal abnormalities
* Surgical complications
* Intraocular lens (IOL) tilt, IOL decentration greater than 0.4 mm (estimated by retroillumination)
* Incomplete follow-up.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sutdy population will be patients implanted bilaterally with the selected multifocal IOL
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
distance,intermediate and near visual acuity | 1, 3 and 6 months

SECONDARY OUTCOMES:
reading speed and contrast sensitivity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcony Santhiago, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Gupta N, Wolffsohn JS, Naroo SA. Comparison of near visual acuity and reading metrics in presbyopia correction. J Cataract Refract Surg. 2009 Aug;35(8):1401-9. doi: 10.1016/j.jcrs.2009.03.026. PMID 19631128
- [Background] Biber JM, Sandoval HP, Trivedi RH, de Castro LE, French JW, Solomon KD. Comparison of the incidence and visual significance of posterior capsule opacification between multifocal spherical, monofocal spherical, and monofocal aspheric intraocular lenses. J Cataract Refract Surg. 2009 Jul;35(7):1234-8. doi: 10.1016/j.jcrs.2009.03.013. PMID 19545814
- [Background] Alfonso JF, Fernandez-Vega L, Amhaz H, Montes-Mico R, Valcarcel B, Ferrer-Blasco T. Visual function after implantation of an aspheric bifocal intraocular lens. J Cataract Refract Surg. 2009 May;35(5):885-92. doi: 10.1016/j.jcrs.2009.01.014. PMID 19393889
- [Background] Hayashi K, Yoshida M, Hayashi H. All-distance visual acuity and contrast visual acuity in eyes with a refractive multifocal intraocular lens with minimal added power. Ophthalmology. 2009 Mar;116(3):401-8. doi: 10.1016/j.ophtha.2008.09.052. Epub 2009 Jan 18. PMID 19152978